CLINICAL TRIAL: NCT02597634
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy, and Safety of SST-0225, a Topical Ibuprofen Cream, in the Treatment of Delayed Onset Muscle Soreness (DOMS)
Brief Title: Study of SST-0225 Topical Ibuprofen Cream in the Treatment of Delayed Onset Muscle Soreness (DOMS)
Acronym: DOMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Strategic Science & Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SST0225-013
Record Dates: First submitted 2015-10-13; First posted 2015-11-05 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Delayed Onset Muscle Soreness, DOMS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SST-0225 (Experimental): Subjects will be treated with IP for 48 hours. While on-site, subjects will apply the first dose of IP at 0 hours, the second dose at 2 hours, and all subsequent doses every 5 (±1) hours, up to a maximum of 6 doses in 24 hours. After subjects complete their 24 hour post first dose NRS pain/soreness on movement assessment, they will be released from the clinic and will continue outpatient treatment for the remaining 24 hours. While off-site subjects will dose every 5 (±1) hours, not to exceed 6 doses in 24 hours.
  Interventions: Drug: SST-0225
- Placebo (Placebo Comparator): Subjects will be treated with IP for 48 hours. While on-site, subjects will apply the first dose of IP at 0 hours, the second dose at 2 hours, and all subsequent doses every 5 (±1) hours, up to a maximum of 6 doses in 24 hours. After subjects complete their 24 hour post first dose NRS pain/soreness on movement assessment, they will be released from the clinic and will continue outpatient treatment for the remaining 24 hours. While off-site subjects will dose every 5 (±1) hours, not to exceed 6 doses in 24 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SST-0225 — SST-0225 is a cream formulation for topical application. Each 5.4 g dose is formulated to topically deliver 400 mg of ibuprofen. The cream contains sodium ibuprofen and various salts.
  Other Names: Topical Ibuprofen Cream
  Arms: SST-0225
Drug: Placebo — Placebo IP will be the same vehicle as SST-0225 vehicle without the active ingredient, ibuprofen. It will be matched in appearance, smell, consistency, and color to SST-0225 topical ibuprofen cream.
  Other Names: Placebo Cream
  Arms: Placebo

SUMMARY:
This is a Phase 3, prospective, randomized, dual-center, double-blind, placebo-controlled, parallel-group study designed to determine the efficacy and safety of SST-0225 (5.4 grams, applied up to 6 times in 24 hours, over a 48-hour dosing period) for the treatment of pain associated with DOMS.

DETAILED DESCRIPTION:
This is a Phase 3, prospective, randomized, multicenter, double blind, placebo controlled, parallel group study designed to determine the efficacy and safety of SST-0225 for the treatment of pain associated with DOMS. Healthy volunteers will be recruited to undergo an exercise regimen designed to induce DOMS in the elbow flexor of the non-dominant arm. Subjects who are eligible following the exercise regimen will be randomized to receive treatment with SST-0225 or placebo for a 48 hour period. Subjects will be housed in the clinic for the first 24 hours of dosing and sent home for the second 24 hour dosing period. Arm pain/soreness will be assessed throughout the study using an 11-point (0-10) Numeric Rating Scale (NRS).

Approximately 150 subjects will be randomized in a 1:1 ratio to SST-0225 or placebo at up to three study centers in the US. Subject participation will be between 12 and 26 days depending on the length of the initial screening period. Once a subject is randomized the duration of participation will be 10 days. The expected duration of the study is approximately six months depending on enrollment. The sample size may be increased to a maximum of 250 based on the results of the planned interim analysis described in Section 15.2 of the protocol.

ELIGIBILITY:
Key Inclusion Criteria The following inclusion criteria will be assessed from the Screening Visit up to the time of randomization:

1. Men and women age 16-65, inclusive
2. Subjects must be able to read, understand, sign, and date the informed consent/assent document indicating they (or a legally acceptable representative) have been informed of all pertinent aspects of the trial
3. Female subjects must agree to use medically acceptable contraceptive methods from the Screening Visit (unless otherwise stated) through end of study (EOS).
4. Subjects must be able to speak, read, and comprehend English or Spanish, and complete required measurements as outlined in the protocol
5. Subjects must agree to refrain from upper body resistance training and any unusual or excessive exercise during the screening period and for the duration of the study, including follow-up
6. Subjects must agree to refrain from the use of restricted therapies during the screening period and until the completion of the dosing period

Key Exclusion Criteria The following exclusion criteria will be assessed from the Screening Visit up to the time of randomization.

1. Subjects who have had an injury to the non-dominant arm such as adhesive capsulitis, bursitis, rotator cuff syndrome, within the six months prior to the Screening Visit
2. Subjects with medial or lateral epicondylitis (tennis elbow) of the non-dominant arm
3. Subjects who have an open wound, skin irritation, or infection on the non-dominant arm in the area to be treated
4. Subjects who have engaged in any upper body resistance training in the six months prior to the Screening Visit
5. Subjects who are actively engaged in manual or physical labor jobs (i.e. brick layer, construction worker, carpenter, house painter)
6. Subjects who should not participate in strenuous exercise for medical reasons
7. Subjects who have abnormal laboratory parameters at the Screening Visit that, in the opinion of the Investigator, could confound interpretation of the study results
8. Subjects with an abnormal physical exam that, in the opinion of the Investigator, would interfere with study participation
9. Subjects who have received oral or injectable systemic corticosteroids within three months prior to the Screening Visit
10. Subjects with osteoarthritis of the hands, fingers, elbows, or shoulders
11. Subjects with chronic pain
12. Subjects with an allergy or a history of allergy or intolerance to aspirin, NSAIDs, acetaminophen or any of the excipients in the IP (L-arginine hydrochloride, glyceryl stearate, cetyl alcohol, squalane, xanthan gum, isopropyl myristate, oleic acid, propylene glycol, polysorbate 20, methyl paraben, phenoxyethanol, propyl paraben, dimethicone)
13. Subjects with current viral or bacterial infections
14. Subjects with certain medical conditions, including:

    1. Peptic ulcer disease
    2. Fibromyalgia
    3. Clinically important gastrointestinal, renal, or hepatic disease within the past six months, in the opinion of the Investigator
    4. Clinically significant cardiovascular disease, in the opinion of the Investigator, not stable for the past six months
    5. Uncontrolled hypertension as indicated by systolic blood pressure ≥ 160 mmHg or a diastolic blood pressure ≥ 100 mmHg
    6. Coagulation disorders or hematologic disease
    7. History of seizures
    8. Known, significant, pre-existing conditions that in the opinion of the Investigator would affect the interpretation of any study data.
15. Subjects with certain myopathies or metabolic defects, including:

    1. Polymyositis (inflammatory)
    2. Sickle cell trait (genetic)
    3. Lipid metabolism disorders (carnitine deficiency, carnitine palmitoyl transferase [CPT] deficiency, β-oxidation enzyme defects)
    4. Glucose metabolism disorders (phosphorylase deficiency [McArdle's Disease], glycolysis enzyme defects).
16. Subjects who have taken anticoagulants, angiotensin-converting enzyme inhibitors, lithium or methotrexate within 30 days prior to the Screening Visit
17. Subjects who are currently taking tricyclic antidepressants including, but not limited to the following:

    1. amitriptyline
    2. clomipramine (Anafranil™)
    3. doxepin (Sinequan®)
    4. imipramine (Tofranil™)
    5. trimipramine (Surmontil®)
    6. amoxapine (Amoxapine Tablets)
    7. desipramine (Norpramin®)
    8. nortriptyline (Pamelor™)
    9. protriptyline (Vivactil®)
18. Subjects with known alcohol abuse, drug dependency, or history of significant psychiatric illness within the past 12 months prior to the Screening Visit
19. Subjects who have used an investigational drug within 30 days prior to the Screening Visit
20. Subjects who are taking diuretics, statins, cyclosporine, or colchicine
21. Subjects with a positive drug screen
22. Females who are pregnant or lactating
23. Subjects who are color-blind

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
SPID24 (calculated by summing the time weighted NRS pain/soreness on movement assessment differences from baseline) | First 24 hours after first dose
  The primary efficacy endpoint will be the time weighted summed pain/soreness intensity difference from baseline NRS pain/soreness on movement assessments over the first 24 hours (SPID24) following the first application of IP on Day 1. SPID24 will be calculated by summing the time weighted NRS pain/soreness on movement assessment differences from baseline (pre-dose on Day 1) to 24 hours (using actual reported NRS assessment times) post first dose of IP on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wade, MD, Principal Investigator — Site #201; David Seiden, MD, Principal Investigator — Site #203; Kayce Morton, DO, Principal Investigator — Site #202
Locations (3):
- United States (3):
  - Site #203, Hollywood, Florida
  - Site #201, South Miami, Florida
  - Site #202, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: Undecided